CLINICAL TRIAL: NCT02293083
Title: Effect of Hyaluronidase Addition to Lidocaine for Trigger Point Injection in Myofascial Pain Syndrome
Brief Title: Hyaluronidase for Trigger Point Injection in Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ji Won Choi, clinical fellowship, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201003046001
Record Dates: First submitted 2014-11-11; First posted 2014-11-18 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Experimental): Group L received trigger point injection with a 3.2 ml of a 1:1 mixture of 1% lidocaine and 0.9% normal saline
  Interventions: Drug: trigger point injection
- Hyaluronidase (Experimental): Group H received trigger point injection with the same volume of solution supplemented with hyaluronidase (H-LASE®, 1500 iu, L&H Pharm., Seoul, Korea) 600 iu/ml
  Interventions: Drug: trigger point injection

INTERVENTIONS:
Drug: trigger point injection

SUMMARY:
Myofascial pain syndrome (MPS) is the most common cause of persistent regional pain characterized by myofascial trigger points. Trigger point injection (TPI) using local anesthetics is one of the most effective methods for treatment of MPS, and steroids or botulinum toxin can be added to local injections .

Recent study suggested that the hyaluronan (HA) could be the basis of myofascial pain. HA within the deep fascia facilitates the free sliding of two adjacent fibrous fascial layers. If the HA assumes a more packed conformation, or more generally, if the loose connective tissue inside the fascia alters its density, the behavior of the entire deep fascia and the underlying muscle would be compromised.

The investigators anticipated that hyaluronidase could decrease the viscosity of HA near the muscle and fascia of trigger points. Meanwhile, hyaluronidase is thought to promote the spread of local anesthetic solution by hydrolyzing glycosidic bonds within HA. Hyaluronidase was shown to be effective in retro- and peribulbar block for ophthalmologic surgery or reducing tissue edema in dermatology, and adhesiolysis for some interventional pain managements.

However, the effect of the addition of hyaluronidase to local anesthetics during TPI has not been studied. The investigators aimed to compare the efficacy of TPI with the addition of hyaluronidase compared to local anesthetic alone on pain and quality of life in MPS patients.

DETAILED DESCRIPTION:
Study approval was obtained from Institutional Review Board (IRB) of Samsung medical center, and written informed consent was obtained from all participants.

The required sample size was determined by power analysis on the basis of a previous study. The primary outcome was pain intensity in the posterior neck and upper back after TPI using verbal numerical rating scale (VNRS). The standard deviation of VNRS was assumed to be 20. Power calculations indicated that detecting 20 points difference in VNRS between the two groups (with α = 0.05 and β = 0.1) would require a sample of 29 subjects for each group. To account for dropouts, 33 subjects were recruited for each group.

Group L received TPI with a 3.2 ml of a 1:1 mixture of 1% lidocaine and 0.9% normal saline. Group H received TPI with the same volume of solution supplemented with hyaluronidase (H-LASE®, 1500 iu, L&H Pharm., Seoul, Korea) 600 iu/ml. The investigators monitored vital sign and any signs of complications such as bleeding, hematoma, allergic reactions for 30 minutes. Treatment efficacy was evaluated by one of the authors (J.W.C.) using VNRS. To reduce bias, this evaluator and the participants were not informed of the assigned group.

Patients' characteristics such as age, height, weight, BMI and pretreatment neck disability index (NDI) and brief pain inventory (BPI) were analyzed by independent t-test. The sex distribution was analyzed by the chi-square test. P values were corrected by Bonferroni's method. Pretreatment VNRS and the duration of pain were evaluated by the Wilcoxon two-sample test. Repeated measures ANOVA was used to compare changes in the VNRS over time between the two groups. Pre- and post-TPI changes in NDI and BPI were compared between the two groups with the Wilcoxon signed rank test and the independent t-test, respectively. All analyses were performed with SPSS 18.0 (SPSS Inc., Chicago, IL, USA) statistical software. Significance was assumed for P values of less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Aged 25-75 years
* Diagnosed with myofascial pain syndrome affecting both trapezius muscles

Exclusion Criteria:

* History of allergy to lidocaine or hyaluronidase
* Anticoagulant medication or antiplatelet agent within 5 days before the study
* Analgesic medication, including non-steroidal anti-inflammatory drugs, tramadol, acetaminophen, or opioids within 5 days of the study
* Pain related to trauma within 6 months before the study
* History of cervical or shoulder surgery
* TPI within 3 months in the same region
* Fibromyalgia
* Cervical radiculopathy or myelopathy
* Obesity, defined as body mass index of 27.5 or higher
* Other medical or psychological conditions (cancer, rheumatoid arthritis, endocrine disease, major depression, schizophrenia)

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Degree of pain as measured by the verbal numerical rating scale | within 2 weeks after intervention